CLINICAL TRIAL: NCT03594370
Title: Multiple Noninvasive Examination Modality to Evaluate the Severity of Ocular Surface Disorders
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201803133RINC
Record Dates: First submitted 2018-07-01; First posted 2018-07-20 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-05

CONDITIONS: Limbal Stem-cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Impression cytology(IC) is a technique which permits the retrieval of the outermost layer of ocular surface cells via the use of various types of filters. It is a minimally invasive method of evaluating human conjunctival epithelial cell morphology. IC may also be utilized in the diagnosis of other ocular diseases, such as ocular surface squamous neoplasia, ocular surface infections, keratoconus and thyroid orbitopathy. IC improves our understanding of the pathophysiology of ocular surface disease, and provide biomarkers to be used as outcome measures in clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control: Limbal image by OCT in normal subjects.
- Advancing wave-like epitheliopathy: Limbal image by OCT in subjects with advancing wave-like epitheliopathy.
- Ocular rosacea or phlyctenulosis: Limbal image by OCT in subjects with ocular rosacea or phlyctenulosis

SUMMARY:
Here the investigators proposed this study to collect cases of different etiologies of ocular surface diseases. With at least one of these four non-invasive examination modalities, the investigators aim to analyze and compare the detecting results. The investigators especially focus on the possibility of using OCT to predict the condition of limbal epithelial stem cells, aiming to use this patient-friendly tool to detect the patient's limbal conditions.

DETAILED DESCRIPTION:
In vivo confocal microscopy, anterior segment optical coherence tomography, keratograph and impression cytology are noninvasive, rapid and easily repeatable technique to investigate ocular surface disorders. In vivo confocal microscopy (IVCM) enables morphological and quantitative analysis of ocular surface microstructure. Optical coherence tomography (OCT) allows for imaging of the morphology of biological tissue with micrometer scale resolution at imaging depths of 1 to 2mm below the tissue surface. [1,2] Anterior segment OCT (ASOCT) has been developed to evaluate corneal diseases[3-8] in different layers. Keratography includes noninvasive meibography and tear interferometry. The former demonstrates the morphology of meibomian glands whereas the later observes quality and quantity of the lipid layer of the tear film. Impression cytology shows the morphology of the corneal and conjunctival epithelial cells, their staining behavior, and nuclear/cytoplasmic ratio could be observed in detail.

Here the investigators proposed this clinical trial to collect cases of different etiologies of ocular surface diseases. With at least one of these four non-invasive examination modalities, the investigators aim to analyze and compare the detecting results. The investigators especially focus on the possibility of using ASOCT to predict the condition of limbal epithelial stem cells, aiming to use this patient-friendly tool to detect the patient's limbal conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is able to understand and cooperate with the examination: aged over 5 years.
* Patient or the legal representative is able to read and sign an informed consent form.
* Patient with one of the diagnosis listed below:

  1. limbal insufficiency
  2. phlyctenulosis
  3. ocular rosacea
  4. ocular graft-versus-host disease (GVHD)
  5. dry eye syndrome (both aqueous deficiency or increased evaporative forms of dry eyes)
  6. other ocular surface diseases (advancing wave-like epitheliopathy, long term use of anti-glaucoma eye drops)

Exclusion Criteria

* Patients who decline to receive any of the non-invasive examinations mentions in this clinical trial.
* Patients younger than 5 years old.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Our study is an institutional observation study recruits otherwise healthy patients aging over 5 years old.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
limbal structural abnormality | assess the OCT limbal image at the baseline
  atypical pattern of limbal Palisade of Vogt detected by OCT comparing to normal subjects

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Study Director — NTUH
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No